CLINICAL TRIAL: NCT03748823
Title: A Phase 3, Randomized, Parallel-Group, Multicenter, Open-Label, Pharmacokinetic, Noninferiority Study of Ravulizumab Administered Subcutaneously Versus Intravenously in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria Currently Treated With Eculizumab
Brief Title: Ravulizumab Subcutaneous (SC) Versus Ravulizumab Intravenous (IV) in Adults With Paroxysmal Nocturnal Hemoglobinuria (PNH) Currently Treated With Eculizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-303; 2017-002370-39 (EudraCT Number)
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Ravulizumab SC Treatment Group (Experimental): In the Randomized Treatment Period, participants will receive an IV loading dose of ravulizumab on Day 1 followed by SC maintenance doses of ravulizumab administered via the ravulizumab OBDS on Day 15 and every week (qw) thereafter for a total of 10 weeks of study treatment.
  In the Extension Period, ravulizumab SC will be administered via the ravulizumab OBDS from Day 71 qw through Day 1274.
  Interventions: Combination Product: Ravulizumab OBDS; Biological: Ravulizumab
- Ravulizumab IV Treatment Group (Active Comparator): In the Randomized Treatment Period, participants will receive an IV loading dose of ravulizumab on Day 1 followed by IV maintenance doses of ravulizumab on Day 15.
  In the Extension Period, ravulizumab SC will be administered via the ravulizumab OBDS from Day 71 qw through Day 1274.
  Interventions: Combination Product: Ravulizumab OBDS; Biological: Ravulizumab

INTERVENTIONS:
Combination Product: Ravulizumab OBDS — The ravulizumab OBDS is a biological-device combination product consisting of a prefilled cartridge containing ravulizumab SC and an on-body injector.
Biological: Ravulizumab — Administered by IV infusion. Ravulizumab IV doses will be based on participant body weight.
  Other Names: ALXN1210

SUMMARY:
The primary objective of this study is to evaluate pharmacokinetics (PK) of ravulizumab administered subcutaneously via an on-body delivery system (OBDS) compared with intravenously administered ravulizumab in adult participants with PNH who are clinically stable on eculizumab for at least 3 months prior to study entry.

DETAILED DESCRIPTION:
The study will consist of up to a 30-day Screening Period, a 10-week Randomized Treatment Period, and an Extension Period of up to 172 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Treated with eculizumab for PNH for at least 3 months prior to Day 1
* LDH level ≤1.5 × upper limit of normal (ULN) at screening
* PNH diagnosis confirmed by documented high-sensitivity flow cytometry.
* Documented meningococcal vaccination not more than 3 years prior to, or at the time of, initiating study treatment.
* Body weight ≥40 to <100 kilogram (kg)
* Female participants of childbearing potential must use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.
* Willing and able to give written informed consent and comply with study visit schedule.

Exclusion Criteria:

* More than 1 LDH value > 2 × ULN within the 3 months prior to study entry
* History of bone marrow transplantation.
* History of or ongoing major cardiac, pulmonary, renal, endocrine, or hepatic disease that, in the opinion of the Investigator or Sponsor, would preclude participation.
* Unstable medical conditions (for example, myocardial ischemia, active gastrointestinal bleed, severe congestive heart failure, anticipated need for major surgery within 6 months of randomization, coexisting chronic anemia unrelated to PNH).
* Females who are pregnant, breastfeeding or who have a positive pregnancy test at screening or Day 1.
* Participation in another interventional clinical study or use of any experimental therapy within 30 days before initiation of study drug on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- Research Site, Los Angeles, California, United States
- Australia (2):
  - Research Site, Liverpool
  - Research Site, Parkville
- Research Site, Vienna, Austria
- Belgium (4):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Hasselt
  - Research Site, Leuven
- Brazil (5):
  - Research Site, Botucatu
  - Research Site, Ribeirão Preto
  - Research Site, Rio de de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
- Research Site, Toronto, Ontario, Canada
- Research Site, Helsinki, Finland
- France (13):
  - Research Site, Amiens
  - Research Site, Brest
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Tours
- Italy (4):
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Roma
  - Research Site, Rome
- Research Site, Maastricht, Netherlands
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg
- Spain (7):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Research Site, Uppsala, Sweden
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Istanbul
  - Research Site, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yenerel MN, Sicre de Fontbrune F, Piatek C, Sahin F, Fureder W, Ortiz S, Ogawa M, Ozol-Godfrey A, Sierra JR, Szer J. Phase 3 Study of Subcutaneous Versus Intravenous Ravulizumab in Eculizumab-Experienced Adult Patients with PNH: Primary Analysis and 1-Year Follow-Up. Adv Ther. 2023 Jan;40(1):211-232. doi: 10.1007/s12325-022-02339-3. Epub 2022 Oct 22. PMID 36272026
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ALXN1210-PNH-303&attachmentIdentifier=429e6f23-2b5d-4a0c-bda6-c3d88e9f946c&fileName=ALXN1210-PNH-303-body_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified by weight group (≥40 to <60 kilogram [kg] and ≥60 to <100 kg) and then randomized in a 2:1 ratio to 2 treatment groups.
Groups:
- Ravulizumab Intravenous (IV)/Subcutaneous (SC) Treatment Group: During the Randomized Treatment Period, participants received a weight-based single loading dose (2400 to 2700 milligrams [mg]) of ravulizumab IV on Day 1, followed by a maintenance weight-based dose (3000 to 3300 mg) of ravulizumab IV on Day 15. During the Extension Period (Day 71 up to Day 1275), participants received 490 mg of ravulizumab SC once every week (qw).
- Ravulizumab SC/SC Treatment Group: During the Randomized Treatment Period, participants received a weight-based single loading dose (2400 to 2700 mg) of ravulizumab SC on Day 1, followed by maintenance weight-based doses (490 mg) of ravulizumab SC qw from Days 15 to 64. During the Extension Period (Day 71 up to Day 1275), participants received 490 mg of ravulizumab SC qw.
Period: Randomized Treatment Period
Arm/Group | Ravulizumab Intravenous (IV)/Subcutaneous (SC) Treatment Group | Ravulizumab SC/SC Treatment Group
Started | 46 | 90
Received at Least 1 Dose of Study Drug | 46 | 90
Treated and Not Included in Analysis (Participants from 1 site with source documentation deviations and findings related to deficiencies in Investigator oversight.) | 1 | 6
Full Analysis Set (Participants who had signed informed consent, randomized, received at least 1 dose of ravulizumab (participants from one noncompliant site were excluded from analysis).) | 45 | 84
Safety Analysis Set (All participants who received at least 1 dose of ravulizumab (participants from one noncompliant site were excluded from analysis).) | 45 | 84
Completed | 44 | 84
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Site Source Document Deviations | 1 | 6
Period: Extension Period
Arm/Group | Ravulizumab Intravenous (IV)/Subcutaneous (SC) Treatment Group | Ravulizumab SC/SC Treatment Group
Started | 44 | 83 (1 participant withdrew consent prior to entering the Extension Period.)
Received at Least 1 Dose of Study Drug | 44 | 83
Treated But Not Included in the Analysis (Participants from 1 site with source documentation deviations and findings related to deficiencies in Investigator oversight.) | 1 | 6
Completed | 31 | 64
Not Completed | 13 | 19
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Death | 2 | 2
Not completed — Other than Specified | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who had signed informed consent, were randomized, received at least 1 dose of ravulizumab, and were not excluded from analysis.
Groups:
- Ravulizumab IV/SC Treatment Group: During the Randomized Treatment Period, participants received a weight-based single loading dose (2400 to 2700 mg) of ravulizumab IV on Day 1, followed by a maintenance weight-based dose (3000 to 3300 mg) of ravulizumab IV on Day 15. During the Extension Period (Day 71 up to Day 1275), participants received 490 mg of ravulizumab SC qw.
- Total: Total of all reporting groups
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group | Total
Number analyzed (Participants) | 45 | 84 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.22) | 45.3 (14.47) | 45.7 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 44 | 69
  Male | 20 | 40 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 15 | 22
  Not Hispanic or Latino | 29 | 53 | 82
  Unknown or Not Reported | 9 | 16 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 29 | 63 | 92
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 7 | 14 | 21

OUTCOME MEASURES:

1. Primary Outcome: Ctrough Serum Concentration of Ravulizumab
Time Frame: Predose at Day 71
Population: Pharmacokinetic (PK) analysis set included all participants who had evaluable PK data.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (µg/mL)
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 43 | 70
micrograms/milliliter (µg/mL) | 457.58 (108.491) | 578.70 (140.819)
Statistical Analysis 1: Comparison: Ravulizumab IV/SC Treatment Group vs Ravulizumab SC/SC Treatment Group; Test type: Non-Inferiority — Noninferiority was determined based on the 90% Confidence interval calculated from the combination z-score that accounts for the interim analysis; p < 0.0001, ANOVA — Analysis of variance (ANOVA) was performed on log-transformed Ctrough and included treatment and stratified weight group as fixed effects; Ratio of Geometric Least Squares Mean = 1.257, 90% CI 2-sided [1.160 to 1.361] — Geometric least squares mean are the least squares mean from the mixed model after back transformation to the original scale. The 90% confidence interval is presented after back transformation to the original scale

2. Secondary Outcome: Ctrough Serum Concentration of Ravulizumab at Day 351
Time Frame: Predose at Day 351
Population: SC treated full analysis set included all participants who had signed informed consent, were randomized, received at least 1 dose of ravulizumab SC, and were not excluded from analysis. Here, Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 34 | 74
µg/mL | 712.79 (203.180) | 737.65 (208.894)

3. Secondary Outcome: Free Serum Complement Component 5 (C5) Concentrations at Day 71
Time Frame: Predose at Day 71
Population: Pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of ravulizumab and who had evaluable PD data. Here, Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 83
µg/mL | 0.072193 (0.0245225) | 0.059458 (0.0182180)

4. Secondary Outcome: Free Serum Complement Component 5 (C5) Concentrations at Day 351
Time Frame: Predose at Day 351
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 33 | 73
µg/mL | 0.071627 (0.0227980) | 0.069711 (0.0208784)

5. Secondary Outcome: Percent Change From Baseline in Lactate Dehydrogenase (LDH) Levels at Day 71
Description: Baseline was defined as the last assessment prior to first study drug dose. LDH samples impacted by tabletop hemolysis were excluded from the analysis.
Time Frame: Baseline, Day 71
Population: Full analysis set included all participants who had signed informed consent, were randomized, received at least 1 dose of ravulizumab, and were not excluded from analysis. Here, Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 43 | 82
percent change | 5.73 (29.716) | 2.57 (33.883)

6. Secondary Outcome: Percent Change From Baseline in LDH Levels at Day 351
Description: SC baseline was defined as the last assessment prior to first dose of SC treatment. LDH samples impacted by tabletop hemolysis were excluded from the analysis.
Time Frame: Baseline, Day 351
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 34 | 73
percent change | -0.83 (17.225) | 1.74 (21.905)

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Subscale Version 4 Score at Day 71
Description: FACIT-fatigue subscale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Items are scored on a 5 point Likert-type scale. Item scores ranged from 0 ("not at all") to 4 ("very much"). The total, summed score ranged from 0 to 52; lower scores indicating greater fatigue and higher score indicating better health-related quality of life. Baseline was defined as the last non-missing value prior to the first dose of study drug.
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 80
units on a scale | -0.83 (7.378) | 1.21 (7.882)

8. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale Version 4 Score at Day 351
Description: FACIT-fatigue subscale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Items are scored on a 5 point Likert-type scale. Item scores ranged from 0 ("not at all") to 4 ("very much"). The total, summed score ranged from 0 to 52; lower scores indicating greater fatigue and higher score indicating better health-related quality of life. Baseline was defined as the last non-missing value prior to the first dose of subcutaneous treatment.
Time Frame: Baseline, Day 351
Population: SC treated full analysis set included all participants who had signed informed consent, were randomized, received at least 1 dose of ravulizumab SC, and were not excluded from analysis. Here, Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure. This outcome measure was planned to be reported for ravulizumab SC/SC treatment group only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 70
units on a scale | 2.57 (7.178)

9. Secondary Outcome: Change From Baseline in Treatment Administration Satisfaction Questionnaire (TASQ) Score at Day 71
Description: The Treatment Administration Satisfaction Questionnaire (TASQ) is a 19-item questionnaire that assesses treatment administration satisfaction across 5 domains: physical impact, psychological impact, impact on activities of daily living, convenience, and satisfaction. Each domain offers up to 5 response options; lower scores indicate a more positive response. Scoring is completed by summing each of the 5 domains. Total TASQ scores during the study ranged from 0 to 367, with a lower score indicating greater satisfaction with treatment administration.
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 43 | 78
units on a scale | -7.00 (34.581) | -70.54 (70.522)

10. Secondary Outcome: Change From Baseline in Treatment Administration Satisfaction Questionnaire (TASQ) Score at Day 351
Description: as for outcome 9
Time Frame: Baseline, Day 351
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 72
units on a scale | -69.29 (80.068)

11. Secondary Outcome: Percentage of Participants Who Experienced Breakthrough Hemolysis up to Day 71
Description: Breakthrough hemolysis was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 grams/deciliter (g/dL)], major adverse vascular event [MAVE, including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2*upper limit of normal (ULN). Denominator for a percentage was participants with at least one post-baseline data for the period. For Through Day 71, only visits with data were used to assess breakthrough hemolysis.
Time Frame: Baseline up to Day 71
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 45 | 84
percentage of participants | 2.2 [0.06 to 11.77] | 1.2 [0.03 to 6.46]

12. Secondary Outcome: Percentage of Participants Who Experienced Breakthrough Hemolysis up to Day 351
Description: Breakthrough hemolysis was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia [hemoglobin <10 g/dL], major adverse vascular event [MAVE, including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH ≥2*ULN. Denominator for a percentage was participants with at least one post-baseline data for the period.
Time Frame: Baseline up to Day 351
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 84
percentage of participants | 4.5 [0.56 to 15.47] | 3.6 [0.74 to 10.08]

13. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Avoidance up to Day 71
Description: Transfusion Avoidance was defined as participants who remained transfusion free and did not require a transfusion after the first dose of study drug through the period of interest. Percentages are based on participants with any post-baseline data for the period. For Through Day 71, only visits with data were used to assess transfusion avoidance.
Time Frame: Baseline up to Day 71
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 45 | 84
percentage of participants | 86.7 [73.21 to 94.95] | 94.0 [86.65 to 98.04]

14. Secondary Outcome: Percentage of Participants Who Achieved Transfusion Avoidance up to Day 351
Description: Transfusion Avoidance was defined as participants who remained transfusion free and did not require a transfusion after the first dose of study drug through the period of interest. Denominator for a percentage was participants with at least one post-baseline data for the period.
Time Frame: Baseline up to Day 351
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 84
percentage of participants | 79.5 [64.70 to 90.20] | 85.7 [76.38 to 92.39]

15. Secondary Outcome: Percentage of Participants Who Maintained Stabilized Hemoglobin (SHg) up to Day 71
Description: SHg was defined as the avoidance of a ≥2 g/dL decrease in hemoglobin level from Baseline (defined as the last assessment prior to the first dose of the study drug) in the absence of transfusion to the end of the period of interest. Percentages were based on participants with at least one post-baseline data for the period. For Through Day 71, only visits with data were used to assess SHg.
Time Frame: Baseline up to Day 71
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 78
percentage of participants | 81.8 [67.29 to 91.81] | 93.6 [85.67 to 97.89]

16. Secondary Outcome: Percentage of Participants Who Maintained SHg up to Day 351
Description: SHg was defined as the avoidance of a ≥2 g/dL decrease in hemoglobin level from SC Baseline (defined as the last assessment prior to the first dose of SC treatment) in the absence of transfusion to the end of the period of interest. Denominator for a percentage was participants with at least one post-baseline data for the period. Visits were based on the number of days since first dose of SC treatment.
Time Frame: Baseline up to Day 351
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
Number analyzed (Participants) | 44 | 79
percentage of participants | 72.7 [57.21 to 85.04] | 83.5 [73.51 to 90.94]

ADVERSE EVENTS:
Time Frame: Baseline up to approximately 3.5 years
Description: Safety analysis set included all participants who received at least 1 dose of ravulizumab and were not excluded from analysis.
Arm/Group | Ravulizumab IV/SC Treatment Group | Ravulizumab SC/SC Treatment Group
All-Cause Mortality (participants affected / at risk) | 2/45 | 2/84
Serious Adverse Events (participants affected / at risk) | 16/45 | 30/84
Other Adverse Events (participants affected / at risk) | 44/45 | 83/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ravulizumab IV/SC Treatment Group (N=45) | Ravulizumab SC/SC Treatment Group (N=84)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lens dislocation (Eye disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Application site induration (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 6
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Tubo-ovarian abscess (Infections and infestations) | 0/25 | 1/44 — This adverse event is gender specific.
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Adnexal torsion (Reproductive system and breast disorders) | 0/25 | 1/44 — This adverse event is gender specific.
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Breakthrough haemolysis (Blood and lymphatic system disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Dengue haemorrhagic fever (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ravulizumab IV/SC Treatment Group (N=45) | Ravulizumab SC/SC Treatment Group (N=84)
Anaemia (Blood and lymphatic system disorders) | 4 | 12
Haemolysis (Blood and lymphatic system disorders) | 4 | 10
Diarrhoea (Gastrointestinal disorders) | 3 | 17
Abdominal pain (Gastrointestinal disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 5 | 9
Vomiting (Gastrointestinal disorders) | 3 | 7
Constipation (Gastrointestinal disorders) | 1 | 6
Pyrexia (General disorders) | 7 | 20
Asthenia (General disorders) | 3 | 13
Influenza like illness (General disorders) | 0 | 7
Injection site erythema (General disorders) | 1 | 7
Fatigue (General disorders) | 3 | 7
Cholelithiasis (Hepatobiliary disorders) | 3 | 4
COVID-19 (Infections and infestations) | 16 | 39
Nasopharyngitis (Infections and infestations) | 8 | 11
Upper respiratory tract infection (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 3 | 11
Influenza (Infections and infestations) | 6 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 7
Headache (Nervous system disorders) | 14 | 16
Dizziness (Nervous system disorders) | 4 | 5
Device delivery system issue (Product Issues) | 42 | 74 — Adverse Events relating to drug delivery were coded to the MedDRA SOC of "Product Issues", including missing dose (ie, no dose) and partial dose (ie, less than full volume of dose administered) medication errors occurring with use of device.
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 6
Toothache (Gastrointestinal disorders) | 4 | 10
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Infusion site erythema (General disorders) | 3 | 4
Gastroenteritis (Infections and infestations) | 5 | 5
Paronychia (Infections and infestations) | 3 | 1
Post vaccination fever (Injury, poisoning and procedural complications) | 4 | 6
Insomnia (Psychiatric disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 1 | 5
Depression (Psychiatric disorders) | 3 | 2
Haemoglobinuria (Renal and urinary disorders) | 3 | 1
Intermenstrual bleeding (Reproductive system and breast disorders) | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
To ensure the quality of the study results, all 7 participants from a noncompliant investigative site were excluded from all prespecified analysis sets due to important source documentation deviations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03748823/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT03748823/SAP_002.pdf